CLINICAL TRIAL: NCT03334513
Title: Refractive and Biometric Outcomes in Patients With Retinopathy of Prematurity Treated With Intravitreal Injection of Ranibizumab as Compared With Bevacizumab - a Clinical Study of Correction at Three Years of Age
Brief Title: Refractive Error and Biometry in Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: San Ni Chen (Other)
Responsible Party: Sponsor-Investigator, San Ni Chen, medical doctor, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Other Study IDs: 171026
Record Dates: First submitted 2017-11-01; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Retinopathy of Prematurity
Keywords: Bevacizumab; Biometry; Ranibizumab; Refractive error; Retinopathy of prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Refractive Errors | interventions — Bevacizumab; Ranibizumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ROP group: children with retinopathy of prematurity received either bevacizumab or ranibizumab
  Interventions: Drug: Bevacizumab; Drug: Ranibizumab

INTERVENTIONS:
Drug: Bevacizumab — intravitreal injection of bevacizumab
  Other Names: avastin
Drug: Ranibizumab — intravitreal injection of ranibizumab
  Other Names: lucentis

SUMMARY:
The investigators compared long-term refractive and biometric outcomes in children with retinopathy of prematurity who received two different anti-vascular endothelial growth factor agents.

DETAILED DESCRIPTION:
Purpose:

To compare refractive and biometric outcomes in patients with type 1 retinopathy of prematurity (ROP) treated with intravitreal injection of Ranibizumab (IVR), versus bevacizumab (IVB), at a corrected age of 3 years.

Methods:

A retrospective case series compared cycloplegic refractive statuses and biometric statuses in patients who received either IVR or IVB for Type 1 ROP, from April 2011 to April 2014.

Comparison of refractive errors and biometric findings between the two groups was performmed and multivariate analysis of possible factors contributive to visual acuity was also performmed

ELIGIBILITY:
Inclusion Criteria:

* children with type 1 retinopathy of prematurity
* children received anti-vascular endothelial growth factors (bevacizumab or ranibizumab)

Exclusion Criteria:

* children withour retinopathy of prematurity
* children with retinopathy of prematurity received laser therapy

Ages: 3 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants who received intravitreal injection of ranibizumab or bevacizumab as the primary treatment
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
spherical equivalent | at corrected age of 3 year-old
  spherical power + half of cylinder power
astigmatism | at corrected age of 3 year-old
  in cylinder power

SECONDARY OUTCOMES:
axial length | at corrected age of 3 year-old
  axial length in mm
cornea radius | at corrected age of 3 year-old
  cornea radius in mm
anterior chamber depth | at corrected age of 3 year-old
  anterior chamber depth in mm
lens thickness | at corrected age of 3 year-old
  lens thickness in mm

REFERENCES:
- [Result] Chen SN, Lian I, Hwang YC, Chen YH, Chang YC, Lee KH, Chuang CC, Wu WC. Intravitreal anti-vascular endothelial growth factor treatment for retinopathy of prematurity: comparison between Ranibizumab and Bevacizumab. Retina. 2015 Apr;35(4):667-74. doi: 10.1097/IAE.0000000000000380. PMID 25462435
- [Derived] Chen YC, Chen SN, Yang BC, Lee KH, Chuang CC, Cheng CY. Refractive and Biometric Outcomes in Patients with Retinopathy of Prematurity Treated with Intravitreal Injection of Ranibizumab as Compared with Bevacizumab: A Clinical Study of Correction at Three Years of Age. J Ophthalmol. 2018 Mar 11;2018:4565216. doi: 10.1155/2018/4565216. eCollection 2018. PMID 29713524